CLINICAL TRIAL: NCT06002243
Title: Non-Expert Acquisition and Remote Expert Review of Screening Echocardiography Images From Child Health and AnteNatal Clinics (NEARER SCAN)
Brief Title: Non-Expert Acquisition & Remote Expert Review of Screening Echocardiography Images From Child Health & AnteNatal Clinics
Acronym: NEARER SCAN
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Menzies School of Health Research (Other)
Collaborators: The University of Western Australia (Other); Telethon Kids Institute (Other); Western Australian Country Health Service (Unknown); Northern Territory Government of Australia (Other Government); Timor-Leste Ministry of Health (Unknown); Miwatj Health Aboriginal Corporation (Unknown); Mala'la Health Service Aboriginal Corporation (Unknown); Pilbara Aboriginal Health Alliance (Unknown)
Responsible Party: Principal Investigator, Joshua Francis, Senior Research Fellow, Menzies School of Health Research
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: APP2015869
Record Dates: First submitted 2023-06-13; First posted 2023-08-21 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Rheumatic Heart Disease
Keywords: Echocardiography; Task-sharing; Aboriginal and Torres Strait Islander Peoples; Pregnancy; Children; First Nation Peoples
MeSH Terms: conditions — Rheumatic Heart Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Participant receiving echocardiography screening.
  Interventions: Diagnostic Test: SPLASH echocardiography screening

INTERVENTIONS:
Diagnostic Test: SPLASH echocardiography screening — Screening echocardiogram performed by a briefly trained health worker with images reviewed off site by an expert cardiologist or cardiac sonographer to determine screening outcome. Screening outcome may include: screen positive, screen negative or uninterpretable images.

SUMMARY:
The Non-Expert Acquisition and Remote Expert Review of Screening echocardiography images from Child health and AnteNatal clinics (NEARER SCAN) study is a co-designed, implementation research project that will improve equitable access to culturally safe, best quality care for Rheumatic Heart Disease (RHD) in high-burden Aboriginal and Torres Strait Islander communities in Australia, and in Timor-Leste. The research addresses an area of unmet need, using novel technologies and embedding them in health practice, to enhance and accelerate diagnosis of RHD outside acute health settings and improve outcomes. The study will be conducted in partnership with community leaders and local partners.

DETAILED DESCRIPTION:
This study titled 'Non-Expert Acquisition and Remote Expert Review of Screening echocardiography images from Child health and AnteNatal clinics' (NEARER SCAN; "LENO BESIK" in Tetum) aims to co-design, implement and evaluate a task-sharing approach to echocardiographic screening for early detection and management of rheumatic heart disease (RHD) in high-risk settings in Australia and Timor-Leste.

Specific objectives include:

1. To co-design implementation strategies with communities underpinned by local program theories.
2. To implement SPLASH echocardiography training and a task-sharing approach to echocardiographic screening for early detection and management of RHD in communities, based on co-designed implementation strategies.
3. To conduct a realist evaluation to understand what implementation strategies assist in integrating this intervention into routine health service delivery and why.
4. To determine the clinical effectiveness of the intervention in terms of impact on key clinical outcome measures.
5. To conduct cost-of-illness, cost-effectiveness and budget-impact analyses of the task-sharing approach to echocardiographic screening for early detection and management of RHD in Australia and Timor-Leste.

Local primary health clinic staff will be trained to perform focused echocardiography using hand-carried ultrasound (HCU) devices employing the 'Single Parasternal Long Axis view with a Sweep of the Heart' (SPLASH) technique. The acquired images will be interpreted by experts (cardiologists and cardiac sonographers) remotely from the site of acquisition. Approximately 1500 children and pregnant women will be screened across high-risk communities in Australia and Timor Leste, over an 18 month period.

A mixed-methods effectiveness-implementation study design will be used to evaluate the implementation of an intervention designed to achieve early detection and management of RHD in high-risk populations. An implementation strategy will be co-designed at each site with the local community and participating primary healthcare (PHC) service, incorporating non-adaptable elements of the intervention, and mapped onto a Theory of Change framework. Co-design, implementation and evaluation will occur simultaneously, and a Type 2 hybrid design study will be used to evaluate both the implementation strategies and the clinical effectiveness of the intervention. The clinical effectiveness will be assessed as the change in the proportion of the at-risk population that received secondary prophylaxis by the end of the study compared to baseline. Program implementation will be evaluated with a realist evaluation to explain under what circumstances the program is successfully integrated into routine service delivery. Data informing evaluation will include numbers of normal, abnormal, and uninterpretable SPLASH echocardiograms obtained, numbers of participants progressing through the cascade of care, augmented by qualitative data from interviews conducted with staff and participants, and costs.

ELIGIBILITY:
Inclusion Criteria in Australia:

* Any child between the age of 5 - 20 years old living in the participating community
* Pregnant women at high risk for RHD undergoing antenatal appointments or a hospital admission will be invited to participate. High risk for RHD will be defined as being from an area where RHD all-age prevalence is >1/1000 RHD or acute rheumatic fever incidence >30/100,000 per year in 5-14-year-olds. For practical purposes, this means Aboriginal women living in urban, rural or remote communities in northern Australia, or immigrants from high-risk settings.

Inclusion criteria for Timor-Leste:

* Any child between the age of 5-20 years old and any pregnant woman.

Exclusion criteria for Australia and Timor-Leste:

* Women who are unable to consent due to physical, mental, or intellectual disability will be excluded. Women and children with known existing cardiac disease will NOT be excluded since evaluation of severity and change in severity during pregnancy will be tracked, and data will inform the calculation of prevalence.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in proportion receiving secondary antibiotic prophylaxis | 18 months from commencement of study
  The change in proportion of the at-risk population receiving secondary antibiotic prophylaxis at the end of the study as compared to baseline

SECONDARY OUTCOMES:
Full echocardiogram following screening echocardiogram | 3 months from screening echocardiogram
  Proportion of people with an abnormal or uninterpretable screening echocardiogram who get a full diagnostic echocardiogram within 3 months and receive a diagnosis.
Proportion of people diagnosed with RHD who are retained in care | 18 months from commencement of study
  Proportion of people diagnosed during study period with RHD who receive guideline-based care by local health service
Secondary antibiotic prophylaxis prescription and adherence | 12 months from time of diagnosis or at end of the study (which ever is longer).
  Proportion of people prescribed secondary prophylaxis who are achieving >= 80% adherence in a 12 months period from time of diagnosis or the end of the study, whichever is longer.
Maternal morbidity and mortality outcomes | Within 6 weeks of the individual's post-partum period
  Description of maternal morbidity and mortality in pregnant women diagnosed with RHD on echocardiographic screening. This will be reported in absolute numbers and percentage of study population. Morbidity will include cardiac complications (heart failure, arrhythmia, aborted sudden cardiac death, acute myocardial infarction), need for obstetric intervention including emergency cesarean section, intensive care admission, other obstetric complications.
Prevalence of rheumatic heart disease within the screened population | 18 months from commencement of study
  Prevalence of RHD in screened population based on echocardiographic diagnosis
Rheumatic valvular heart disease severity (mild, moderate or severe) within the screening population based on echocardiographic diagnosis | 18 months from commencement of study
  Description of severity of RHD in screened population. This will include proportions of mild, moderate and severe valve disease.
Neonatal morbidity and mortality outcomes | Within 6 weeks post-partum
  Description of neonatal morbidity and mortality outcomes for the pregnant women diagnosed with RHD. This will be reported as absolute numbers and percentage of study population. Morbidity will include need for admission to neonatal intensive care.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua R Francis, MBBS, Principal Investigator — Menzies School of Health Research

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jones B, Marangou J, Yan J, Ralph A, Mitchell A, Kaethner A, Remenyi B, Wade V, Katzenellenbogen JM, Monteiro AF, Cannon JW, Howard NJ, Gilles M, Haynes E, Seixas H, Maurays J, Neave J, Pears C, Engelman D, Canuto K, Steer A, Unger H, Bailey M, Tanesi M, Amaral S, Neto H, Stewart M, Burgess P, Brown A, Currie BJ, Hillis G, Morris P, Simon D, Wheaton G, Williamson J, de Dassel J, Slota-Kan S, Carapetis J, English M, Nagraj S, Francis JR. NEARER SCAN (LENO BESIK) evaluation of a task-sharing echocardiographic active case finding programme for rheumatic heart disease in Australia and Timor-Leste: protocol for a hybrid type II effectiveness-implementation study. BMJ Open. 2024 Oct 18;14(10):e083467. doi: 10.1136/bmjopen-2023-083467. PMID 39424380